CLINICAL TRIAL: NCT04713215
Title: Thinking Outside the Box: Exploring Patient and Carer Perceptions of Medication Compliance Aids (MCAs)
Brief Title: Thinking Outside the Box
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other); Sir Halley Stewart Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: 289976; 2782 (Other Grant/Funding Number: Sir Halley Stewart Trust)
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2021-07

CONDITIONS: Medication Compliance; Medication Adherence; Caregivers; Attitude
Keywords: Medication Compliance; Medication Adherence; Caregivers; Attitude
MeSH Terms: conditions — Medication Adherence; Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Patients where MCAs are currently being used: Intervention: Patient questionnaire - Part A - patients where MCAs are currently being used
  Interventions: Other: Questionnaire
- Patients where an MCA was discontinued: Intervention: Patient questionnaire - Part B - patients where an MCA was discontinued
  Interventions: Other: Questionnaire
- Patients where an MCA was declined: Intervention: Patient questionnaire - Part C - patients where an MCA was declined
  Interventions: Other: Questionnaire
- Carers where MCAs are currently being used: Intervention: Carer questionnaire - Part A - carers where MCAs are currently being used
  Interventions: Other: Questionnaire
- Carers where an MCA was discontinued: Intervention: Carer questionnaire - Part B - carers where an MCA was discontinued
  Interventions: Other: Questionnaire
- Carers where an MCA was declined: Intervention: Carer questionnaire - Part C - carers where an MCA was declined
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A short (approximately 20-minute) questionnaire will be administered to patients and carers who meet the inclusion criteria and who have expressed and interested, and consented to completing the questionnaire.

SUMMARY:
Medication adherence - the extent to which a patient takes their medications as prescribed - is a global problem. Half of all medicines given to patients with long-term health problems are not taken properly by the patient. Older adults are also more at risk of harm from their medications as they tend to take more medicines than young people, and are less able to cope with their effects.

There has been research into how to address these problems. One way has been through providing patients with a medication compliance aid (MCA), to help with taking their medications on time. MCAs are pre-packaged boxes containing tablets, grouped together according to the day and time the medication needs to be taken. Some patients buy the MCA and fill it themselves, other patients collect a MCA that their pharmacy makes for them.

There is not much proof that pharmacy-filled MCAs help patients, and some research suggests they may cause harm. The views of patients on MCA use have not yet been fully explored - it is not clear why some patients choose to stop using an MCA or refuse one when offered. Many patients with MCAs also have a family member or friend who helps them with their medication. No research has recognised the role of informal carers in helping patients with MCAs or asked them their thoughts.

This study aims to understand what patients, aged 65 and older, and their informal carers think about MCAs and how they affect their lives. It is a questionnaire study which will take place within a National Health Service (NHS) hospital. It's designed to take approximately 20 minutes, either face to face or by phone. The investigators hope that the results from this study will help to inform how healthcare professionals use MCAs to the benefit of patients and their carers.

DETAILED DESCRIPTION:
Definitions Patient is defined as a service user in a hospital/outpatient/community setting, who may or may not have used an MCA in the past.

Informal Carer is a person who, in an unpaid capacity, supports a Patient in some aspect of their care - for the scope of this study, this must include assistance with medication. They will also be referred to as a Carer. It must be noted that paid carers are outside the scope of this study. A paid carer is someone in formal employment in a caring capacity.

Participant is defined as either a Patient or Informal Carer who consents to be part of the study, and have their data stored and used for the purposes outlined in this protocol.

Medication Compliance Aid(s), also referred to as Medication Aid(s) or MCAs, are pre-packaged boxes containing tablets correctly grouped together according to the day and time the medication needs to be taken, assembled by a pharmacist.

Research participants for this study will belong to the following 4 groups:

1. Patients (inpatient or outpatient) aged 65 or over currently using an MCA
2. Patients (inpatient or outpatient) aged 65 or over previously offered an MCA but declined/discontinued
3. Informal carers (aged 18 or over) of patients (aged 65 or over) using MCAs.
4. Informal carers (aged 18 or over) of patients (aged 65 or over) who were previously offered an MCA but it was declined/discontinued

All participants must be able to speak English and have sufficient cognitive function to provide informed consent.

Patients and informal carers will not be recruited in pairs (i.e patient and their informal carer). The investigators will be recruiting informal carers of patients that have cognitive impairment and some of the patients with cognitive impairment will not have sufficient capacity to partake in the survey themselves. However, their informal carers are an important and large group of those supporting patients with their medications and therefore need to be included in this study.

Setting:

Data collection for this single-centre study will be taken from participants identified through various means including outpatient attendees (telephone and face to face), inpatient wards and community settings e.g. a hospital @home team. The hospital @home team involves a "community ward", involving doctors, nurses, pharmacists and therapy teams employed by the same NHS Foundation Trust, where clinicians assess and treat patients in their homes.

Informal carers who assist with medications are identified in these settings as part of normal clinical practice on hospital admission, clinic or @home review and also in discharge planning activities.

The investigators will also place posters in an outpatient clinic waiting room within the older persons assessment unit, to advertise the study to patients and informal carers.

Identification of participants:

Potential participants will be approached and screened by their clinical care team during the course of routine clinical activity. A member of the direct clinical team will approach potential participants, confirm eligibility using a standardised set of screening questions, describe the study briefly and ask for verbal consent for their name and phone number to be passed to the research team. Informal carers are commonly identified by clinical teams as part of routine admission questions when a patient is admitted to hospital, as formal (paid) care arrangements need to be distinguished from informal arrangements for the purpose of discharge assessment and onward care at home. Identification of who assists with the patient's medications is also identified as part of routine care by pharmacy staff. The investigators will encourage members of the direct clinical care team to ask informal carers the screening questions during routine care discussions and whether they would be interested in taking part. If yes, the clinical team member will pass on their contact details.

If a patient lacks capacity to give informed consent for inclusion in the study, they will not be approached for participation. Informal carers of these patients who meet the informal carer inclusion criteria will still be eligible to be approached and will be contacted by the clinical team looking after the patient in the first instance to check eligibility and inquire regarding whether they are interested in taking part. This contact will be during a routine clinical activity such as obtaining a collateral history from an informal carer.

Recruitment: On approach by researcher, participants will be given a description of the study verbally (face to face or via phone). All potential participants will be given a copy of the written participant information sheet prior to completing the questionnaire.

Verbal consent to proceed with the questionnaire will be sought. Optional consent will also be sought to record a participant's email or postal address to disseminate a lay summary of results on completion of the study.

Questionnaire:

Participants will complete a short questionnaire containing a mix of quantitative and qualitative questions with scope to include free-text comments.

The questions will vary according to whether the participant is a patient or carer, and whether they are currently using a pharmacy-filled MCA, previously discontinued a pharmacy-filled MCA or have previously declined a pharmacy-filled MCA. The questions will explore the following;

For patients, and the informal carers of patients, who use MCAs

1. Establish patient and informal carer opinions of MCAs
2. Determine whether those who use MCAs would consider switching to taking medicines in their original packaging

For patients, and the informal carers of patients, who have used an MCA in the past but no longer do so

1. Establish patient and informal carer opinions of an MCA
2. Explore patient and informal carers reasons for stopping an MCA
3. Explore alternative ways in which patients and informal carers organise medications without the use of an MCA

For patients and their informal carers who have been offered an MCA but declined

1. Explore why the MCA was declined
2. Explore alternative ways in which patients and their informal carers organise medications without the use of an MCA
3. To explore what further support they would like to help them adhere to their medications

The researchers will administer the questionnaire in all settings including face to face and phone call. This will broaden participation to those who have difficulty reading and writing.

Close of interaction:

The participant will be thanked for their time and any further questions will be answered. No further interactions will occur.

ELIGIBILITY:
Patient inclusion criteria:

* Patients currently using an MCA or patients previously offered an MCA but declined or discontinued
* Age 65 years or older
* English speaker
* Sufficient cognitive function to complete questionnaire

Informal Carer inclusion criteria:

* A person who cares for someone aged 65 or older who is currently using a MCA or previously offered an MCA and declined or discontinued
* They assist the person they care for with their medication.
* Age 18 years or older
* English speaking
* Sufficient cognitive function to complete questionnaire

Patient exclusion criteria:

* Age less than 65 years
* Lacks capacity to consent to participate in study
* Deemed by the direct clinical care team to be too unwell to participate
* Declines participation

Informal carer exclusion criteria:

* Age less than 18 years
* Employed to assist patient
* Not involved with medication management
* Lacks capacity to consent to participate in study
* Declines participation

All participants must be able to speak English and have sufficient cognitive function to provide informed consent. Patients and carers will not all be recruited in pairs (i.e a patient and their carer). If a patient lacks capacity to give informed consent for inclusion in the study, they will not be approached for participation. Informal carers of these patients who meet the informal carer inclusion criteria will still be eligible to be approached.

Ages: 18 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Patients aged 65 or over currently using an MCA
  * Patients aged 65 or over previously offered an MCA but discontinued
  * Patients aged 65 or over previously offered an MCA but declined
  * Informal carers (aged 18 or over) of patients aged 65 or over, currently using an MCA
  * Informal carers (aged 18 or over) of patients aged 65 or over, who were previously offered an MCA but discontinued
  * Informal carers (aged 18 or over) of patients aged 65 or over, who were previously offered an MCA but declined
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
To determine patients' and carers' opinions of medication compliance aids | 12 months
  Through qualitative and quantitative analysis

SECONDARY OUTCOMES:
To determine whether those using MCAs would consider reverting to medicines in original packaging and what they might require to support this change. | 12 months
  Through qualitative and quantitative analysis

CONTACTS AND LOCATIONS:
Overall Officials: Rebekah Schiff, BSc, MBBS, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thielemans L, Chin K, Hegarty A, Schiff R. Carer involvement in medication adherence: carer views and experiences of facilitating medication adherence using pharmacy-filled multi-compartment medication compliance aids and other methods of adherence support-a questionnaire survey. Age Ageing. 2023 Oct 2;52(10):afad169. doi: 10.1093/ageing/afad169. PMID 37930740